CLINICAL TRIAL: NCT05206292
Title: Estimating Prevalence of Inherited Disorders of Sulfur Amino Acids Metabolism in Patients With Psychotic Disorders.
Acronym: PsyNIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC21.0294; 2021-A01940-41 (Other: ID RCB)
Record Dates: First submitted 2022-01-06; First posted 2022-01-25 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Inherited Metabolic Disorder of Nervous System; Schizophrenia
Keywords: NIT1; Sulfitest; Inherited Metabolic Disorder; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Adult patients with psychotic disorder without known organic cause.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient cohort (Other): There is only one patient arm. It corresponds to the cohort of included patients, all of whom had psychotic disorders with no known organic etiology.
  Interventions: Diagnostic Test: Sulfitest

INTERVENTIONS:
Diagnostic Test: Sulfitest — Urine strip to detect the presence of sulfites in urine. Immediate result.

SUMMARY:
Screening for sulfur amino acid metabolism pathologies using a sulfitest in adult patients with psychotic disorder.

DETAILED DESCRIPTION:
Psychotic disorder is a public health problem, with a cumulative incidence in the general population estimated at 3%. Although in most cases the origin is purely psychiatric, psychotic disorder can also represent a mode of entry into many organic pathologies. Among these, hereditary metabolic diseases, although rare in the general population, hold a special place, especially in view of their potentially treatable character. However, the identification of this type of disease within the mass of patients with psychotic disorders can be an extremely complex task, and has been the subject of scientific interest for many years.

Recently, at the Grenoble Alpes University Hospital, a new hereditary metabolic disease that causes psychotic disorders has been discovered. This disease was identified in a family of patients, most of whom had psychotic disorders, and all of whom had deep cystic leukoencephalopathy on MRI and a positive sulfitest. The discovery of this new hereditary metabolic disease raises the question of its prevalence in patients with psychotic disorders, and more generally of the prevalence of diseases of sulfur amino acid metabolism.

PsyNIT study therefore aims, using the sulfitest, to detect hereditary diseases of sulfur amino acid metabolism in a sample of patients with psychotic disorders without known organic etiology. The discovery of other patients would raise the question of screening more widely for this type of pathology, and would modify the management of the patients thus screened in terms of follow-up and possibly treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older,
* Followed for a psychotic disorder,
* With no known organic etiology for the psychotic disorder,
* Not having formulated its opposition to participation in the study (or his/her tutor/curator),
* Affiliated with the social security system.

Exclusion Criteria:

* Patients protected by law (minors, pregnant or breastfeeding women, deprived of liberty or hospitalized under constraint, under administrative or judicial supervision) except patients under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of positive sulfitests (compared to the number of patients included). | 15 minutes
  Sulfitest is considered positive if clearly colored.

SECONDARY OUTCOMES:
Sulfite concentration in urine (semi-quantitative scale). | 15 minutes
  Sulfite concentration is estimated by visual analysis of the urine dipstick test.
Clinical characteristics of patients with a positive sulfitest. | 15 minutes
  Collection of clinical characteristics of patients with a positive sulfitest, by questioning or by analysis of the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Besson, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perala J, Suvisaari J, Saarni SI, Kuoppasalmi K, Isometsa E, Pirkola S, Partonen T, Tuulio-Henriksson A, Hintikka J, Kieseppa T, Harkanen T, Koskinen S, Lonnqvist J. Lifetime prevalence of psychotic and bipolar I disorders in a general population. Arch Gen Psychiatry. 2007 Jan;64(1):19-28. doi: 10.1001/archpsyc.64.1.19. PMID 17199051
- [Result] Sedel F, Baumann N, Turpin JC, Lyon-Caen O, Saudubray JM, Cohen D. Psychiatric manifestations revealing inborn errors of metabolism in adolescents and adults. J Inherit Metab Dis. 2007 Oct;30(5):631-41. doi: 10.1007/s10545-007-0661-4. Epub 2007 Aug 10. PMID 17694356
- [Result] Rendu J, Van Noolen L, Garrel C, Brocard J, Marty I, Corne C, Faure J, Besson G. Familial deep cavitating state with a glutathione metabolism defect. Ann Clin Transl Neurol. 2019 Dec;6(12):2573-2578. doi: 10.1002/acn3.50933. Epub 2019 Nov 9. PMID 31705625
- [Result] Peracchi A, Veiga-da-Cunha M, Kuhara T, Ellens KW, Paczia N, Stroobant V, Seliga AK, Marlaire S, Jaisson S, Bommer GT, Sun J, Huebner K, Linster CL, Cooper AJL, Van Schaftingen E. Nit1 is a metabolite repair enzyme that hydrolyzes deaminated glutathione. Proc Natl Acad Sci U S A. 2017 Apr 18;114(16):E3233-E3242. doi: 10.1073/pnas.1613736114. Epub 2017 Apr 3. PMID 28373563
- [Result] Misko AL, Liang Y, Kohl JB, Eichler F. Delineating the phenotypic spectrum of sulfite oxidase and molybdenum cofactor deficiency. Neurol Genet. 2020 Jul 14;6(4):e486. doi: 10.1212/NXG.0000000000000486. eCollection 2020 Aug. PMID 32802950